CLINICAL TRIAL: NCT03032276
Title: Impact and Operational Assessment of an Integrated Safe Motherhood and Newborn Health Promotion Package: a Community-based Cluster Randomized Controlled Trial
Brief Title: Safe Motherhood Promotion and Newborn Survival
Acronym: SMPNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Government of Bangladesh (Other Government); Tokyo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-16013
Record Dates: First submitted 2017-01-11; First posted 2017-01-26 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2021-12

CONDITIONS: Neonatal Death; Maternal Death
Keywords: Safe motherhood; Newborn survival; Community; Cluster Randomized Trial
MeSH Terms: conditions — Perinatal Death; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): "'Safe motherhood and newborn health promotion package'" will be implemented in the intervention arm which comprise 15 randomly selected unions (lowest level of administrative unit).
  Interventions: Other: Safe motherhood and newborn health promotion package
- Comparison (No Intervention): Another 15 union will be selected where no intervention will be implemented

INTERVENTIONS:
Other: Safe motherhood and newborn health promotion package — The intervention package consists of three components: facility, community and linkages between the community and health facilities. Facility based interventions will serve both the comparison and intervention arms. However, other two interventions will serve the intervention arm only. Specific interventions and approaches for the three components will be implemented within the MOH&FW service delivery system to improve MNH practices in families and communities and to increase the use of MNH services from appropriate facilities/providers. The intervention package has been developed based on the experiences from SMPP in Narsingdi district and on the basis of consultations with the International Advisory Body (IAB) that included GoB, JICA, ICDDR,B, other experts and stakeholders.
  Arms: Intervention

SUMMARY:
Primary objective of the study is to measure the impact of a comprehensive package of interventions introduced by the Safe Motherhood Promotion and Newborn Survival project on neonatal mortality in three Upazila of Chandpur district, Bangladesh

DETAILED DESCRIPTION:
Burden: Globally around 6.3 million children under five years of age died in 2013, two third of which occur in the low & middle income countries. Bangladesh is one of the LMICs countries with high burden of maternal and neonatal mortalities. In Bangladesh, there has been a considerable progress in reduction of both child and maternal mortality in recent decades. From 1994 to 2014 under-5 mortality rate has reduced from 133 to 46 per 1000 live births in Bangladesh; however, within the same timeframe neonatal mortality declined from 52 to 28 per 1000 live births. This slow decrease in newborn deaths means that it now constitutes a greater share of total under-5 deaths. At present, neonatal mortality accounts for 74% of deaths in infants and 61% in children aged less than 5 years. Similarly, the country was able to decline MMR by 70% between 1990 and 2013, from 574 to 170 per 100,000 live births, with an annual reduction rate of 5.0%. Such statistics highlights the importance of focusing on perinatal and early postnatal periods to prevent maternal and neonatal mortalities.

Knowledge gap: Safe motherhood promotion project (SMPP) was a five (5 yr) year pilot project, launched in July 2006, by the Government of Bangladesh (GOB) in collaboration with JICA. The aim of the project was to improve the health status of pregnant and postpartum women and neonates. SMPP implemented three linked activities i.e., advocacy at the central level, strengthening of health facilities and empowerment of community. Evaluation of SMPP found positive changes in UN process indicators on EmOC including met needs (up from 31% to 55%), case fatality rate (<0.1%) and skilled birth attendance rate (from 18% to 25%). The major weakness of the previous assessment of SMPP were use of a before-after design without any concurrent comparison area and the assessment lacked population based mortality estimates, only measured hospital case fatality rate. Hence, there is lack of strong evidences regarding the impact of the project.

Relevance: The proposed project is expected to provide essential evidences to the GOB and other development partners with the help of stronger design and valid evaluation processes. It would help not only in prioritizing, planning, and further scaling-up of SMPNS interventions in other areas of Bangladesh but in informing other developing countries in similar settings also.

Hypothesis: Safe Motherhood and Newborn Survival intervention package will reduce neonatal mortality by 25%, in comparison to the routine services in Chandpur district, Bangladesh

Methods: A community-based, cluster-randomized design will be used to evaluate the effectiveness of an integrated "Safe Motherhood and Newborn Health Promotion Package" in Chandpur district, Bangladesh. Both quantitative and qualitative approaches will be employed to address the primary and secondary objectives. Baseline, midterm and end of intervention household survey will be conducted using validated structured questionnaire to assess the coverage of maternal & newborn health interventions. Health facility assessments surveys will be conducted periodically to assess facility readiness and utilization of maternal and neonatal health services in the participating health facilities. Additionally, relevant data from routine Health Management Information System (HMIS) will be regularly collected and extracted An ongoing investigating system will be in place at the health facilities to identify and document maternal near miss cases.

Qualitative data will be collected for process documentation and in depth exploration of implementation challenges and contextual factors. Social capitals will be measured both quantitatively and qualitatively to assess the non health impact of the interventions. Qualitative data collection methods will include stakeholders' meeting, focus group discussions (FGD), periodic in-depth assessments, social mapping and other participatory exercises.

Outcome measures/variables: The primary outcome measure for evaluation of SMPNS intervention is reduction of neonatal mortality. In addition, changes in coverage and utilization of maternal & newborn health services, cost effectiveness of implementation of intervention will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Women with birth outcome in last three years

Exclusion Criteria:

* Unusual unions as per the contextual factors (demographics, terrain, functionality of health services, etc.) will be excluded.
* If a union has a total population of less than 12,000 (the minimum required to get adequate sample of neonates) they will either be excluded

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50400 (Estimated)
Dates: Start 2016-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of neonatal mortality rate (NMR) | During baseline at year 1, in two mid-line at year 2 & 3 and finally after completion of the of the intervention at year 4
  NMR will be assessed at the beginning of the project. after that it will also assessed by two midline assessment after starting the intervention and finally it will be assessed during the endline survey

SECONDARY OUTCOMES:
Changes in coverage and utilization of maternal and newborn health services | At year 1 (baseline), year 2 and 3 (mid lines) and year 4 (end line)
  This will be assessed to evaluate the effect of the comprehensive package of interventions on health and care seeking behavior for neonates and women during antepartum, intrapartum and postpartum period at baseline and end line survey on total population and during two mid line surveys in a sub set of population
Cost effectiveness of implementing the interventions | Every six months for programme costs
  Costs for improved neonatal health outcomes and related health services. This will be assessed by analyzing Costs per DALY averted, Costs per life-year gained; Costs per case of delivery by skilled attendance; Costs per case of essential neonatal care, Program cost, both start up and post implementation, Incremental health service costs for providing quality services, Out of pocket expenditure etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shams El Arifeen, DrPH, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; D M Emdadul Hoque, MPH, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Sanwarul Bari, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Masum Billah, MPH, BURP, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Ahmed Ehsanur Rahman, MPH, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Tazeen Tahsina, MS Economics, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Mohiuddin Ahsanul Kabir Chowdhury, MPH, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Mohammad Mehedi Hasan, MPH, MSc, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Sajia Islam, MPH, BDS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Mohammad Masudur Rahman, MPS, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Nazia Binte Ali, MPH, MBBS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Jasmin Khan, MPH, MSS, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Caulfield LE, de Onis M, Blossner M, Black RE. Undernutrition as an underlying cause of child deaths associated with diarrhea, pneumonia, malaria, and measles. Am J Clin Nutr. 2004 Jul;80(1):193-8. doi: 10.1093/ajcn/80.1.193. PMID 15213048
- [Background] Jones G, Steketee RW, Black RE, Bhutta ZA, Morris SS; Bellagio Child Survival Study Group. How many child deaths can we prevent this year? Lancet. 2003 Jul 5;362(9377):65-71. doi: 10.1016/S0140-6736(03)13811-1. PMID 12853204
- [Background] Victora CG, Wagstaff A, Schellenberg JA, Gwatkin D, Claeson M, Habicht JP. Applying an equity lens to child health and mortality: more of the same is not enough. Lancet. 2003 Jul 19;362(9379):233-41. doi: 10.1016/S0140-6736(03)13917-7. PMID 12885488
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Terra de Souza AC, Peterson KE, Andrade FM, Gardner J, Ascherio A. Circumstances of post-neonatal deaths in Ceara, Northeast Brazil: mothers' health care-seeking behaviors during their infants' fatal illness. Soc Sci Med. 2000 Dec;51(11):1675-93. doi: 10.1016/s0277-9536(00)00100-3. PMID 11072887
- [Background] Baqui AH, Arifeen SE, Williams EK, Ahmed S, Mannan I, Rahman SM, Begum N, Seraji HR, Winch PJ, Santosham M, Black RE, Darmstadt GL. Effectiveness of home-based management of newborn infections by community health workers in rural Bangladesh. Pediatr Infect Dis J. 2009 Apr;28(4):304-10. doi: 10.1097/INF.0b013e31819069e8. PMID 19289979
- [Background] Wakefield SE, Poland B. Family, friend or foe? Critical reflections on the relevance and role of social capital in health promotion and community development. Soc Sci Med. 2005 Jun;60(12):2819-32. doi: 10.1016/j.socscimed.2004.11.012. Epub 2004 Dec 24. PMID 15820589
- [Background] Hawe P, Shiell A. Social capital and health promotion: a review. Soc Sci Med. 2000 Sep;51(6):871-85. doi: 10.1016/s0277-9536(00)00067-8. PMID 10972431
- [Background] Pagel C, Prost A, Lewycka S, Das S, Colbourn T, Mahapatra R, Azad K, Costello A, Osrin D. Intracluster correlation coefficients and coefficients of variation for perinatal outcomes from five cluster-randomised controlled trials in low and middle-income countries: results and methodological implications. Trials. 2011 Jun 14;12:151. doi: 10.1186/1745-6215-12-151. PMID 21672223
- [Background] De Silva MJ, Harpham T, Tuan T, Bartolini R, Penny ME, Huttly SR. Psychometric and cognitive validation of a social capital measurement tool in Peru and Vietnam. Soc Sci Med. 2006 Feb;62(4):941-53. doi: 10.1016/j.socscimed.2005.06.050. Epub 2005 Aug 10. PMID 16095787
- [Background] Bland JM, Altman DG. Cronbach's alpha. BMJ. 1997 Feb 22;314(7080):572. doi: 10.1136/bmj.314.7080.572. No abstract available. PMID 9055718
- [Background] El Arifeen S, Hill K, Ahsan KZ, Jamil K, Nahar Q, Streatfield PK. Maternal mortality in Bangladesh: a Countdown to 2015 country case study. Lancet. 2014 Oct 11;384(9951):1366-74. doi: 10.1016/S0140-6736(14)60955-7. Epub 2014 Jun 29. PMID 24990814
- [Derived] Hoque DME, Chowdhury MAK, Rahman AE, Billah SM, Bari S, Tahsina T, Hasan MM, Islam S, Islam T, Mori R, Arifeen SE. A community-based cluster randomized controlled trial (cRCT) to evaluate the impact and operational assessment of "safe motherhood and newborn health promotion package": study protocol. BMC Public Health. 2018 May 3;18(1):592. doi: 10.1186/s12889-018-5478-6. PMID 29724194